CLINICAL TRIAL: NCT07048613
Title: Comparative Study of Magnetic Resonance Imaging and Transrectal Ultrasound in Identifying Clinically Significant Prostate Cancer Among Diverse Ethnic Groups Using Histopathology as the Gold Standard
Brief Title: Comparative Study of MRI and TU in Identifying Clinically Significant Prostate Cancer Among Ethnic Groups
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/901
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI (mpMRI)
  Interventions: Diagnostic Test: MRI (mpMRI)

INTERVENTIONS:
Diagnostic Test: MRI (mpMRI) — : Combines T2-weighted imaging, Diffusion-weighted imaging (DWI), and Dynamic contrast-enhanced MRI (DCE-MRI) to provide detailed anatomical images and assess tissue characteristics.

SUMMARY:
This study is designed to compare the diagnostic accuracy of Magnetic Resonance Imaging (MRI) and Transrectal Ultrasound (TRUS) in detecting clinically significant prostate cancer, using histopathology (biopsy results) as the gold standard. Prostate cancer is a leading cause of cancer-related morbidity among men globally, and its detection often varies across ethnic groups due to genetic, environmental, and healthcare access factors. This research aims to evaluate how MRI and TRUS perform across diverse ethnic populations to determine the most reliable imaging modality for early diagnosis.

DETAILED DESCRIPTION:
The study will follow an observational, cross-sectional design. Patients suspected of having prostate cancer will undergo both MRI and TRUS imaging before a prostate biopsy. Imaging findings will be recorded and compared to the histopathological outcomes from biopsy samples. Sensitivity, specificity, positive predictive value, and negative predictive value will be calculated for each modality. Additionally, subgroup analysis will be performed to evaluate performance variations across different ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Male patients who are 40 years of age or older
* Individuals who exhibit increased PSA values (e.g., PSA >4 ng/mL) or abnormal results on a digital rectal examination (DRE), which are clinical indicators of prostate cancer) 16

Exclusion Criteria:

* Individuals who have previously had treatment for prostate cancer, such as hormone therapy, chemotherapy, radiation, or surgery
* Severe comorbidities that make safe imaging or biopsy impossible, such as severe heart failure or end-stage renal disease

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary condition under investigation in this study is clinically significant prostate cancer, a malignant disease affecting the prostate gland in men. The study focuses on the diagnostic evaluation and detection of this condition using two commonly employed imaging techniques: Magnetic Resonance Imaging (MRI) and Transrectal Ultrasound (TRUS).
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | 12 Months
  The EORTC QLQ-C30 is a 30-item questionnaire used to assess the quality of life (QoL) of cancer patients. It consists of five functional scales, three symptom scales, a global health status/QoL scale, and six single-item symptom scales. Scoring involves calculating the average of items within each scale, then linearly transforming the scores to a 0-100 range, with higher scores generally indicating better functioning or higher symptom burden

CONTACTS AND LOCATIONS:
Locations (1):
- Aznostics The Diagnostic Center, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No